CLINICAL TRIAL: NCT07148076
Title: "Perception, Knowledge, and Attitudes of Educational Staff Regarding the Care of Children With Type 1 Diabetes: Evaluation of the Educational Program"
Acronym: PKA-T1D-EDU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sibenik University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Nevena Simunic, Principal Investigator, Lecturer, MSN, Sibenik University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SibenikU
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 Diabetes, Children, Educational Staff, Primary Schools,Kindergartens
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Education Program (Experimental): Participants in the intervention group completed a baseline questionnaire assessing perceptions, knowledge, and attitudes about type 1 diabetes care. They then participated in an educational program specifically designed to improve these aspects. Immediately following the education, participants completed a second questionnaire. A third questionnaire was administered 3 months after the intervention to assess retention of knowledge and changes in attitudes and perceptions.
  Interventions: Behavioral: Education Program
- Control Group - No Intervention (No Intervention): Participants in the control group did not receive any educational program or intervention. They completed the same questionnaire as the intervention group at baseline and again 3 months later. This allowed for comparison of changes in perceptions, knowledge, and attitudes about type 1 diabetes care without exposure to the educational intervention.

INTERVENTIONS:
Behavioral: Education Program — This intervention consists of a structured educational program specifically designed for educational staff in primary schools and kindergartens, focusing on the care of children with type 1 diabetes. The program includes interactive lectures, practical workshops, and case studies covering diabetes management, symptom recognition, emergency procedures, and day-to-day support for children with type 1 diabetes in educational settings. Unlike standard informational sessions or general health education, this intervention is tailored to address the unique challenges and responsibilities faced by school and kindergarten staff. The program is delivered in-person by certified diabetes educators and includes pre- and post-training assessments to measure changes in knowledge, perceptions, and attitudes. Participants are tracked using unique codes to allow for longitudinal comparison of results before, immediately after, and three months following the intervention.
  Arms: Intervention Group - Education Program

SUMMARY:
Type 1 diabetes is a chronic autoimmune disease that requires continuous monitoring and regulation of glycemia. Children with type 1 diabetes face challenges that can disrupt their daily routines in school and kindergarten. This includes the need for self-monitoring, continuous blood sugar measurement, insulin administration, proper nutrition, regular physical activity, and timely interventions in cases of hypoglycemia or hyperglycemia. Therefore, children with diabetes often require support from educational staff, including teachers, preschool educators, and other professional personnel while attending educational institutions.

A safe and supportive (pre)school environment is crucial for maintaining the health and well-being of children with type 1 diabetes. Teachers and preschool educators, as key actors in the daily (pre)school life of the child, play an important role in recognizing disease symptoms and managing emergencies. However, research shows that many teachers lack sufficient knowledge about the symptoms of diabetes and the necessary procedures in emergencies, which can endanger the health and safety of the child, as well as their equal participation in educational activities.

ELIGIBILITY:
Inclusion Criteria:

* Educational staff employed in primary schools and/or kindergartens within the study area
* Individuals willing to participate who have provided informed consent
* Participants available for all planned assessments during the study period.

Exclusion Criteria:

* Educational staff who have type 1 diabetes themselves, to avoid bias in the assessment of knowledge, perceptions, and attitudes due to personal experience with the disease
* Educational staff who have close family members (parent, child, spouse, sibling) diagnosed with type 1 diabetes, as personal experiences and additional knowledge gained through family circumstances could affect the objectivity of the results
* Individuals unable to participate in all phases of the study (e.g., due to planned absence or other reasons)
* Individuals who are unwilling or unable to provide informed consent
* This description clearly defines who is eligible and who is excluded from participation, ensuring the representativeness and objectivity of the study sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in the perception, knowledge, and attitudes of educational staff regarding the care of children with type 1 diabetes | Before the educational program Immediately after the educational program The entire study is scheduled to be conducted over a period of 10 months
  Primary Outcome:
  The primary outcome will be assessed by measuring the difference in the total score on a comprehensive, structured questionnaire designed to evaluate the perception, knowledge, and attitudes of educational staff regarding the care of children with type 1 diabetes. The questionnaire is administered before and immediately after participation in the educational program, as well as three months post-intervention. The objective is to quantify the immediate and sustained effects of the intervention on participants' understanding and preparedness to support children with type 1 diabetes in educational settings.
  Time Frame:
  Assessment will be conducted at three time points: prior to the start of the educational program (baseline) immediately after completion of the program.
  Instrument:
  The instrument used is a structured questionnaire specifically developed for this study. It is a compilation of seven previously validated instruments

SECONDARY OUTCOMES:
Sustainability of Changes in Knowledge, Perception, and Attitudes | Three months after completion of the educational program
  This outcome will assess the sustainability of changes in educational staff's knowledge, perceptions, and attitudes regarding the care of children with type 1 diabetes. The difference in total scores on the same structured questionnaire will be measured three months after the educational program, compared to both baseline and immediate post-intervention results. This analysis aims to determine whether the improvements observed immediately after the intervention are maintained over time, indicating lasting impact of the educational program on participants' competencies and attitudes.
  Instrument:
  The same structured questionnaire developed specifically for this study, which is a compilation of seven previously validated instruments covering all relevant aspects of diabetes care in educational settings. This tool has undergone expert review and pilot testing to ensure its validity and reliability within the target population.

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - Osnovna škola Tin Ujević, Dječji vrtići Smilje, Šibenik, Hrvatska
  - Osnovna škola Tin Ujević, Dječji vrtići Smilje, Šibenik, Hrvatska 22000, Šibenik, Šibenik

IPD SHARING:
Plan to Share IPD: Undecided